CLINICAL TRIAL: NCT01922921
Title: Phase I/II Randomized Study of Combination Immunotherapy With or Without Polysaccharide Krestin (PSK®) Concurrently With a HER2 ICD Peptide-Based Vaccine in Patients With Stage IV Breast Cancer Receiving HER2-Targeted Monoclonal Antibody Therapy
Brief Title: Vaccine Therapy With or Without Polysaccharide-K in Patients With Stage IV HER2 Positive Breast Cancer Receiving HER2-Targeted Monoclonal Antibody Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, William Rayford Gwin III, MD, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7866; NCI-2013-01377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 135; 7866/135; 7866 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); U19AT006028 (NIH)
Record Dates: First submitted 2013-08-01; First posted 2013-08-14 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: HER2/Neu Positive; Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; 2C4 antibody; polysaccharide-K; Glycoproteins; Trastuzumab; PF-05280014

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (placebo) (Active Comparator): Patients receive HER2 ICD peptide-based vaccine ID once monthly for 3 months, trastuzumab (or trastuzumab and pertuzumab) per standard of care, and placebo PO BID for 4 months.
  Interventions: Biological: HER-2/neu Intracellular Domain Protein; Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Other: Placebo; Biological: Trastuzumab
- Arm II (polysaccharide-K) (Experimental): Patients receive HER2 ICD peptide-based vaccine ID and trastuzumab (or trastuzumab and pertuzumab) as in Arm I and polysaccharide-K PO BID for 4 months.
  Interventions: Biological: HER-2/neu Intracellular Domain Protein; Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Biological: Polysaccharide-K; Biological: Trastuzumab

INTERVENTIONS:
Biological: HER-2/neu Intracellular Domain Protein — Given ID
  Other Names: HER-2 ICD Peptide; HER-2/neu ICD Protein; HER2 ICD; HER2 Intracellular Domain
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pertuzumab — Given per standard of care
  Other Names: 2C4; 2C4 Antibody; MoAb 2C4; Monoclonal Antibody 2C4; Perjeta; rhuMAb2C4; RO4368451
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I (placebo)
Biological: Polysaccharide-K — Given PO
  Other Names: Glycoproteins; Krestin; KS-2; PSK
  Arms: Arm II (polysaccharide-K)
Biological: Trastuzumab — Given per standard of care
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014

SUMMARY:
This randomized phase I/II trial studies the side effects of vaccine therapy with or without polysaccharide-K and to see how well it works in treating patients with stage IV human epidermal growth factor receptor 2 (HER2) positive breast cancer who are receiving HER2-targeted monoclonal antibody therapy. Vaccines made from HER2 intracellular domain (ICD) peptide may help the body build an effective immune response to kill tumor cells that express HER2. Polysaccharide-K may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether vaccine therapy works better when given with or without polysaccharide-K in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of polysaccharide-K (PSK) when given with HER2-directed immunotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the effect of PSK on natural killer (NK) cell functional activity when given with HER2-directed immunotherapy.

TERTIARY OBJECTIVES:

I. To investigate the effect of PSK when given with HER2-directed immunotherapy on: serum levels of pro-inflammatory cytokine and/or chemokines; intermolecular epitope spreading; serum transforming growth factor (TGF)-beta levels; progression free survival (PFS) and overall survival (OS).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive HER2 ICD peptide-based vaccine intradermally (ID) once monthly for 3 months, trastuzumab (or trastuzumab and pertuzumab) per standard of care, and placebo orally (PO) twice daily (BID) for 4 months.

ARM II: Patients receive HER2 ICD peptide-based vaccine ID and trastuzumab (or trastuzumab and pertuzumab) as in Arm I and polysaccharide-K PO BID for 4 months.

After completion of study treatment, patients are followed up for 9 months and then twice annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV HER2+ breast cancer treated to:

  * No evidence of disease (NED), or
  * Stable bone only disease after definitive therapy
* HER2 overexpression by immunohistochemistry (IHC) of 2+ or 3+ in the primary tumor or metastasis; or documented gene amplification by fluorescent in situ hybridization (FISH) analysis; IHC =< 2+ must have HER2 gene amplification documented by FISH
* Patients must continue HER2-targeted monoclonal antibody therapy dosing per standard of care through the entire study period (one year)

  * HER2-targeted monoclonal antibody therapy is defined as either trastuzumab monotherapy, or trastuzumab and pertuzumab combination therapy administered per standard of care
* Patients must be at least 21 days post cytotoxic chemotherapy prior to enrollment
* Patients must be at least 28 days post immunosuppressants prior to enrollment
* Patients must be at least 28 days from use of any mushroom supplements (examples: turkey tail, reishi, maitake, shiitake) and agree to withhold them for the entire study period (one year)
* Patients on bisphosphonates and/or endocrine therapy are eligible
* Patients who are having sex that could lead to pregnancy must agree to contraceptive use during the entire study period
* Patients must have Zubrod performance status score of =< 2
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have significant active concurrent medical illnesses precluding study treatment
* White blood cell (WBC) >= 3000/mm^3
* Hemoglobin (Hgb) >= 10 g/dl
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min
* Total bilirubin =< 1.5 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 times the upper limit of normal
* Patients must have adequate cardiac function as demonstrated by normal left ventricular ejection fraction (LVEF) >= the lower limit of normal for the facility on multi gated acquisition (MUGA) scan or echocardiogram (ECHO) within 3 months of enrollment

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Restrictive cardiomyopathy
  * Unstable angina within 6 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure
  * Symptomatic pericardial effusion
* Patients with any contraindication to receiving rhu granulocyte macrophage colony stimulating factor (rhuGM-CSF) based products
* Patients with any clinically significant autoimmune disease requiring active treatment
* Patients receiving any concurrent immunosuppressants
* Patients who are pregnant or breast-feeding
* Patients who are simultaneously enrolled in other treatment studies
* Patients who have received a previous HER2 breast cancer vaccine
* Known hypersensitivity reaction to mushroom products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lupe Salazar, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Placebo) | Arm II (Polysaccharide-K)
Started | 16 | 15
Completed | 15 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Placebo) | Arm II (Polysaccharide-K) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Median (Full Range); unit: years] | 52 [36 to 62] | 59 [33 to 75] | 52 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 13 | 29
  Italy | 0 | 1 | 1
  Canada | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3 or Higher Toxicity Per Study Arm.
Description: Evaluated using physical examinations and clinical labs by type and grade of toxicities noted during treatment, There were graded per Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events 4.0.
Time Frame: Up to 4 months
Population: Only 1 patient of the 2 patients listed below had a possibly related event of vomiting.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Placebo) | Arm II (Polysaccharide-K)
Number analyzed (Participants) | 16 | 15
Participants | 2 | 0

2. Secondary Outcome: Induction of Interferon (IFN)-Gamma Production and Cluster of Differentiation (CD)107a Expression in NK Cells, Via Flow Cytometry
Description: Augmentation of NK cell activity is defined by a 2-fold increase (at time of maximal change) in NK cell IFN-gamma production and CD107a expression
  For the results we used CD56 which is the accepted phenotypic marker for natural killer (NK) cells and CD16 which is a receptor on NK cells that facilitates antibody-dependent cellular cytotoxicity (ADCC). CD56dim are typically responsible for cytolytic activity and targets cell killing, whereas, CD56bright are the main source of cytokine production (i.e. IFN-gamma). CD56dim CD16bright NK cells represent at least 90% of all peripheral blood NK cells with a maximum of 10% as CD56bright NK cells
  We compared the baseline expression of CD56brightCD16dim or CD56dimCD16bright (prior to start of study treatment) to the maximum expression of CD56brightCD16dim or CD56dimCD16bright at 1 of 4 timepoints after the start of the oral administration of study treatment (polysaccharide-K/placebo (either week 4, 8, 12 or 16).
Time Frame: Up to 16 weeks
Population: Only 9/15 patients were evaluable for this analysis in Arm 1. Only 13/14 patients we evaluable for this analysis in Arm 2.
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Placebo) - CD56dim CD16bright; Arm I (Placebo) - CD56bright CD16dim: Patients receive HER2 ICD peptide-based vaccine ID once monthly for 3 months, trastuzumab (or trastuzumab and pertuzumab) per standard of care, and placebo PO BID for 4 months.
  HER-2/neu Intracellular Domain Protein: Given ID
  Laboratory Biomarker Analysis: Correlative studies
  Pertuzumab: Given per standard of care
  Placebo: Given PO
  Trastuzumab: Given per standard of care
- Arm II (Polysaccharide-K) - CD56dim CD16bright; Arm II (Polysaccharide-K) - CD56bright CD16dim: Patients receive HER2 ICD peptide-based vaccine ID and trastuzumab (or trastuzumab and pertuzumab) as in Arm I and polysaccharide-K PO BID for 4 months.
  HER-2/neu Intracellular Domain Protein: Given ID
  Laboratory Biomarker Analysis: Correlative studies
  Pertuzumab: Given per standard of care
  Polysaccharide-K: Given PO
  Trastuzumab: Given per standard of care
Arm/Group | Arm I (Placebo) - CD56dim CD16bright | Arm II (Polysaccharide-K) - CD56dim CD16bright | Arm I (Placebo) - CD56bright CD16dim | Arm II (Polysaccharide-K) - CD56bright CD16dim
Number analyzed (Participants) | 9 | 13 | 9 | 13
Participants
  INF gamma+: >=2 fold increase | 4 | 9 | 4 | 7
  INF gamma+: <2 fold increase | 5 | 4 | 5 | 6
  CD107+: >=2 fold increase | 3 | 8 | 3 | 6
  CD107+: <2 fold increase | 6 | 5 | 6 | 7

3. Other Pre Specified Outcome: Change in Intermolecular Epitope Spreading Assessed by IFN-gamma Enzyme-linked Immunosorbent Spot Assay
Description: IFN-γ ELISPOT assay will be used to evaluate T cell precursor frequency to specific breast tumor antigens. A positive immune response will be defined as a post-vaccination T cell precursor frequency >1:20,000 antigen-specific PBMCs. In patients with a baseline precursor frequency >1:20,000, a positive post-vaccination immune response will be defined as a 2-fold increase in antigen-specific PBMC. PBMC will be cryopreserved and subsequently be thawed at time of analysis.
Time Frame: Baseline to 12 months after completion of treatment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Pro-inflammatory Serum Cytokine and/or Chemokines Assessed by Luminex Analysis
Time Frame: Baseline to 24 hours after completion of treatment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Serum TGF-beta Levels Assessed by Enzyme-linked Immunosorbent Assay
Time Frame: Baseline to 12 months after completion of treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: OS
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PFS
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Clinical and/or chemical parameters for all study patients will be evaluated for potential toxicity at baseline, before each vaccine, and 1 month after the third vaccine (total of 4 months evaluation).
Description: Toxicity grading will be evaluated per CTEP CTCAE 4.0 and monitoring of AEs will be done per FDA and NCI guidelines. AEs will be tabulated per CTCAE 4.0 system organ class and descriptive statistics will be used to summarize toxicity profiles for the PSK and placebo groups.
Arm/Group | Arm I (Placebo) | Arm II (Polysaccharide-K)
All-Cause Mortality (participants affected / at risk) | 1/16 | 2/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 16/16 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Placebo) (N=16) | Arm II (Polysaccharide-K) (N=15)
Lymphocyte count decreased (Investigations) | 6 (7) | 4 (5) — 4/7 events reported were related to placebo arm 4/5 events reported were related to the treatment arm
White blood cell decreased (Investigations) | 3 (4) | 3 (3) — 4/4 events reported were related to the placebo arm 1/3 events reported were related to the treatment arm
Platelet count decreased (Investigations) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) — 1/1 events reported was related to placebo arm 1/1 events reported was related to the treatment arm
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — 1/1 events reported was related to placebo arm
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — 1/1 events reported was related to placebo arm
Other - rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Anemia (Blood and lymphatic system disorders) | 4 (4) | 6 (7) — 1/4 events reported were related to placebo arm 1/6 events reported were related to treatment arm
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Other - pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Headache (Nervous system disorders) | 1 (1) | 7 (9) — 1/1 events reported was related to placebo arm 6/9 events reported were related to the treatment arm
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 6 (8) — 1/4 events reported were related to placebo arm 7/8 events reported were related to treatment arm
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0) — 3/5 events reported were related to placebo arm
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0) — 2/4 events reported were related to placebo arm
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) — 1/2 events reported were related to placebo arm
Other - minor acid reflux after drinking tea for half hour or so (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0) — 1/3 events reported were related to placebo arm
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Other - acne/rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (6) | 2 (2) — 2/2 events reported were related to the treatment arm
Flu like symptoms (General disorders) | 7 (8) | 7 (12) — 5/8 events reported were related to placebo arm 12/12 events reported were related to treatment arm
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) — 1/1 reported events was related to the treatment arm
Injection site reaction (General disorders) | 14 (29) | 13 (26) — 29/29 events reported were related to placebo arm 25/26 events reported were related to treatment arm
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (2) — 1/1 events reported was related to placebo arm 1/2 events reported were related to treatment arm
Other - head sweats-daily (Vascular disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) — 1/1 reported events was related to treatment arm
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — 1/2 events reported were related to placebo arm
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) — 2/3 events reported were related to treatment arm
Other - dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Other - engorged breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Other - hyperactive-increase senstivity of allergens-food, pollen, bug bite (Immune system disorders) | 1 (1) | 0 (0) — 1/1 events reported was related to placebo arm
Blood bilirubin increase (Investigations) | 0 (0) | 1 (1)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right knee pain increased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left lip cold sores (Herpes) (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Hematochezia - 2 episodes (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) — 3/3 events reported were related to the treatment arm
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) — 1/1 events reported was related to the treatment arm
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Umbilical follicitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scalp skin nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Infusion related reactions (General disorders) | 0 (0) | 1 (1) — 1/1 events reported was related to treatment arm
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — 1/2 events reported were related to the treatment arm
Cystitis - UTI (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT01922921/Prot_SAP_000.pdf